CLINICAL TRIAL: NCT02326103
Title: Randomised Open-label Multicenter Study Evaluating Ciprofloxacin in Severe Alcoholic Hepatitis in Addition to Prednisolon Therapy
Brief Title: Randomised Open-label Multicenter Study Evaluating Ciprofloxacin in Severe Alcoholic Hepatitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Markku Nissinen, chief specialist, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELSINKIU
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Alcoholic Hepatitis; Alcoholic Cirrhosis
Keywords: alcoholic; hepatitis; cirrhosis; cholesterol metabolites; ciprofloxacin
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Cirrhosis, Alcoholic; Hepatitis; Fibrosis | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciprofloxacin (Active Comparator): Oral administration of Ciprofloxacin 500mg twice daily
  Interventions: Drug: Ciprofloxacin
- Placebo (Placebo Comparator): Oral administration of Placebo pill twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin — Comparison of ciprofloxacin with placebo in alcoholic hepatitis
  Arms: Ciprofloxacin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study is aimed to evaluate the additional role of ciprofloxacin therapy in severe alcoholic hepatitis combined to prednisolone therapy in an open-label placebo controlled manner.

DETAILED DESCRIPTION:
Introduction: Alcoholic hepatitis (AH) is an inflammatory liver injury associated with longstanding excess alcohol consumption. Disease spectrum varies from asymptomatic transaminase elevations to fulminate liver failure. In hospital mortality in patients with severe alcoholic hepatitis not responding to corticosteroids is over 30 %.

Alcohol increases gut permeability and promotes the translocation of lipopolysaccharide (LPS) from the gut lumen the portal vein, and further to Kupffer cells, where LPS binds to CD14, ultimately activating multiple cytokine genes.

Diagnosis of AH is based on history of heavy alcohol use, symptoms like jaundice and on typical laboratory findings, and in uncertain cases on liver biopsy.

Determination of the severity of alcoholic hepatitis is essential for assessment of the disease prognosis and selection therapy. Cessation of alcohol consumption is mandatory for further therapy. Several scoring systems are available to assess the severity and the prognosis of alcohol hepatitis. Maddrey discrimination function (DF) is most widely used and enables to identify patients with severe alcohol hepatitis responding to corticosteroid therapy.

The first line therapy in severe alcoholic hepatitis (DF≥32) is prednisolone. However, those not responding to steroids have 77 % 6 months mortality.

New treatment options for severe AH are desperately needed. Although increased bacterial and LPS translocation are considered to have central role in the pathogenesis of AH no controlled studies of antibiotics in alcoholic hepatitis has been published. In Finland 600 AH requiring hospitalization are diagnosed annually.

Study objective: To evaluate to additional role of ciprofloxacin therapy in severe alcoholic hepatitis combined to prednisolone therapy.

Moreover, we try to find new and better predictors for liver injury and treatment response.

Patients: 150 AH patients, with Maddrey DF >32.

Randomization: Patients with severe AH are randomized at hospitalization 1:1 to receive:

1. Prednisolone 40 mg/day for 1 month, with decreasing by 5 mg/week + ciprofloxacin 1000 mg/ day for 120 days or
2. Prednisolone 40 mg/day for 1 month, with decreasing by 5 mg/week + placebo/ day for 120 days Measurement of response Early change in bilirubin levels (ECBL= S-Bil(Day 0)-S-Bil(Day7 )>0 Lille Score >0.45 day 7. Change in serum sterol levels as surrogate markers of cholesterol synthesis (reflecting liver function and severity of cholestasis) Primary end point Mortality at day 28, at 6 months and at 12 months Secondary end points: Proportion of patients with early change in bilirubin levels (ECBL= S-Bil(Day 0)-S-Bil(Day7 )>0 Proportion of patients with Lille Score >0.45 day 7 Recovery of liver function parameters in 1 and 3 months

ELIGIBILITY:
Inclusion Criteria:

Severe alcoholic hepatitis; Maddrey above 300

Exclusion Criteria:

Viral hepatitis Remarkable bleeding in the gastrointestinal tract Serious bacterial infection Hepatorenal syndrome Earlier participation in this study Malignant disease not in remission Other liver disease affecting remarkably the outcome of alcoholic liver disease Mental retardation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Death at 28 days | 28 days after randomisation
Death at 3 months | 3 months after randomisation
Death at 6 months | 6 months after randomisation

SECONDARY OUTCOMES:
Early reduction in serum bilirubin level | 7 days after randomisation
Surrogate markers of liver function | 7 days to 12 months
  Improvement of surrogate markers of cholesterol synthesis and liver synthesis capacity, e.g., lathosterol, cholestenol and desmosterol

CONTACTS AND LOCATIONS:
Overall Officials: Perttu Sahlman, MD, Principal Investigator — University Hospital of Helsinki
Locations (1):
- University Hospital of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers during the study or during the analysis of the results.